CLINICAL TRIAL: NCT02579564
Title: Systemic Chemotherapy Combined With Thoracic Cavity Perfusion of Recombinant Human Adenovirus Type 5 and Endostatin Injections Versus Cisplatin for Treatment Malignant Hydrothorax in Non Small Cell Lung Cancer (NSCLC) Patients: A Multi-center, Randomized, Controlled Clinical Trial
Brief Title: Systemic Chemotherapy Combined With Recombinant Human Adenovirus Type 5 and Endostatin Injections for Treatment Malignant Hydrothorax in NSCLC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Zhengtang Chen, Chief Physician, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTAEMTF
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Malignant Hydrothorax; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Vinorelbine; Paclitaxel; Pemetrexed; endostar protein; Endostatins; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chemotherapy with Oncorine and Endostar (Experimental): Systemic chemotherapy with standard schemes, such as GP (Gemcitabine/Cisplatin), NP (Vinorelbine/Cisplatin), TP (Paclitaxel/Cisplatin) or PP (Pemetrexed/Cisplatin). Thoracic cavity perfusion of recombinant human adenovirus type 5 injection 1.5ml and Endostar 30mg each time, twice a week for four times.
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Oncorine; Drug: Endostar; Drug: Cisplatin
- chemotherapy with cisplatin (Active Comparator): Systemic chemotherapy with standard schemes without cisplatin, such as Gemcitabine, Vinorelbine, Paclitaxel or Pemetrexed. Thoracic cavity perfusion of cisplatin 30mg/m2 each time, twice a week for four times.
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: Vinorelbine
Drug: Paclitaxel
Drug: Pemetrexed
Drug: Oncorine
  Other Names: recombinant human adenovirus type 5 injection
  Arms: chemotherapy with Oncorine and Endostar
Drug: Endostar
  Other Names: recombinant human endostatin injection
  Arms: chemotherapy with Oncorine and Endostar
Drug: Cisplatin

SUMMARY:
The purpose of this multi-center clinical trial is to verify more effective on local control of malignant pleural effusions in NSCLC patients by thoracic cavity perfusion of recombinant human adenovirus type 5 injection and recombinant human Endostatin injection (Endostar) compared with cisplatin perfusion, with acceptable side effects.

DETAILED DESCRIPTION:
Malignant pleural effusion, which can malfunction of circulatory and respiratory systems, is a common complication in advanced NSCLC, finally decreases the quality of life and lifespan. Nowadays, it is still a challenge to effectively control malignant pleural effusion. In this multi-center randomized and controlled clinical trial, 134 NSCLC patients diagnosed as malignant pleural effusion in the first time will enroll. Based on systemic chemotherapy and pleural cavity perfusion, all eligible patients are randomly assigned into treatment group (recombinant human adenovirus type 5 and Endostatin injections) and control group (cisplatin) with ratio 1:1. Local control rate and side effects are record respectively. The anticipation is that treatment group obtains faster and longer control of pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 yrs;
2. Kamofsky score (KPS) ≥70, and a predicted lifespan >3 months;
3. Enough function of vital organs, such as heart, liver and kidney;
4. Advanced NSCLC diagnosed by cytology or pathology
5. Unilateral or bilateral of malignant pleural effusion in the first time;
6. Patients who are considered as malignant pleural effusion by cytology or biomarkers (CEA, CA199, CA125) in pleural effusion;
7. Without systemic infection or high fever;
8. Without active EGFR mutation or unwilling to targeted molecular therapy;
9. NO Anti tumor Radiotherapy chemotherapy and molecular targeted therapy,or Received Anti tumor Radiotherapy chemotherapy and molecular and clinical remission more than three months and in the past month ,disease progress with pleural cavity effusion but haven't use systemic or local anti tumor treatment.
10. No pleural cavity injection of antineoplastic drugs.

Exclusion Criteria:

1. Non-malignant pleural effusion;
2. Pleural effusion cause by other malignant tumors;
3. Allergic to Recombinant human adenovirus type 5 injection or Endostar;
4. Pregnant or lactation women;
5. Previously using Medicine for treating NSCLC with pleural cavity effusion by Systemic or pleural cavity perfusion treatment one month prior to enrollment;
6. Previously using the diuretics, albumin and anti-angiogenesis drugs, or dexamethasone one month prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of malignant pleural effusions | up to 3 years
  Assessed by WHO Cancerous effusion scoring system

SECONDARY OUTCOMES:
progression-free survival | up to 3 years

OTHER OUTCOMES:
quality of life | up to 3 years
  Assessed by Karnofsky Performance Status(KPS)
side effects | up to 3 years
  Assessed by NCI CTC3.0